CLINICAL TRIAL: NCT03107988
Title: Phase 1 Study of Lorlatinib (PF-06463922), an Oral Small Molecule Inhibitor of ALK/ROS1, for Patients With ALK-Driven Relapsed or Refractory Neuroblastoma
Brief Title: NANT 2015-02: A Phase 1 Study of Lorlatinib (PF-06463922)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Approaches to Neuroblastoma Therapy Consortium (Other)
Collaborators: Pfizer (Industry); University of Southern California (Other); Solving Kids' Cancer US/EU (Unknown); Children's Neuroblastoma Cancer Foundation (Unknown); The Band of Parents (Unknown); The Evan Foundation (Other); Wade's Army (Unknown); Ronan Thompson Foundation (Unknown); The Catherine Elizabeth Blair Memorial Foundation (Unknown); Cookies for Kids' Cancer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NANT2015-02
Record Dates: First submitted 2017-03-21; First posted 2017-04-11 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — lorlatinib; Cyclophosphamide; Topotecan; Filgrastim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Cohort A1 DL1 (Experimental): Lorlatinib will be given orally once daily continuously for 28 days. The dose level of lorlatinib will be 45 mg/m2/dose. Patients must be under 18 years of age at time of enrollment.
  Interventions: Drug: Lorlatinib
- Cohort A2 DL 3A (Experimental): Lorlatinib will be given at 100 mg orally once daily continuously for 28 days. Patients must be 18 years of age or older at time of enrollment.
  Interventions: Drug: Lorlatinib
- Cohort B2 DL4B (Experimental): Lorlatinib will be given orally once daily continuously for 28 days at 95mg/m2/dose. Lorlatinib should be administered at least one hour prior to conventional chemotherapy (Cyclophosphamide and Topotecan) on days 1-5 of each cycle. Patients must be under 18 years of age at time of enrollment.
  Interventions: Drug: Lorlatinib; Drug: Cyclophosphamide; Drug: Topotecan; Drug: Filgrastim/pegfilgrastim
- Cohort A1 DL2 (Experimental): Lorlatinib will be given orally once daily continuously for 28 days. The dose level of lorlatinib will be 60 mg/m2/dose. Patients must be under 18 years of age at time of enrollment.
  Interventions: Drug: Lorlatinib
- Cohort A1 DL3 (Experimental): Lorlatinib will be given orally once daily continuously for 28 days. The dose level of lorlatinib will be 75 mg/m2/dose. Patients must be under 18 years of age at time of enrollment.
  Interventions: Drug: Lorlatinib
- Cohort A1 DL4 (Experimental): Lorlatinib will be given orally once daily continuously for 28 days. The dose level of lorlatinib will be 95 mg/m2/dose. Patients must be under 18 years of age at time of enrollment.
  Interventions: Drug: Lorlatinib
- Cohort A1 DL5 (Experimental): Lorlatinib will be given orally once daily continuously for 28 days. The dose level of lorlatinib will be 115 mg/m2/dose. Patients must be under 18 years of age at time of enrollment.
  Interventions: Drug: Lorlatinib
- Cohort A2 DL4A (Experimental): Lorlatinib will be given at 150 mg orally once daily continuously for 28 days. Patients must be 18 years of age or older at time of enrollment.
  Interventions: Drug: Lorlatinib
- Cohort B2 DL5B (Experimental): Lorlatinib will be given orally once daily continuously for 28 days at 115mg/m2/dose. Lorlatinib should be administered at least one hour prior to conventional chemotherapy (Cyclophosphamide and Topotecan) on days 1-5 of each cycle. Patients must be under 18 years of age at time of enrollment.
  Interventions: Drug: Lorlatinib; Drug: Cyclophosphamide; Drug: Topotecan; Drug: Filgrastim/pegfilgrastim
- Cohort B2 DL3A (Experimental): Lorlatinib will be given orally once daily continuously for 28 days at 100mg/day. Lorlatinib should be administered at least one hour prior to conventional chemotherapy (Cyclophosphamide and Topotecan) on days 1-5 of each cycle. Patients must be 18 years of age or older at time of enrollment.
  Interventions: Drug: Lorlatinib; Drug: Cyclophosphamide; Drug: Topotecan; Drug: Filgrastim/pegfilgrastim
- Cohort B2 DL4A (Experimental): Lorlatinib will be given orally once daily continuously for 28 days at 150mg/day. Lorlatinib should be administered at least one hour prior to conventional chemotherapy (Cyclophosphamide and Topotecan) on days 1-5 of each cycle. Patients must be 18 years of age or older at time of enrollment.
  Interventions: Drug: Lorlatinib; Drug: Cyclophosphamide; Drug: Topotecan; Drug: Filgrastim/pegfilgrastim
- Cohort B1 DL5 (Experimental): Lorlatinib will be given orally once daily continuously for 28 days. The dose level of lorlatinib will be 115 mg/m2/dose. Patients must be under 18 years of age at time of enrollment.
  Interventions: Drug: Lorlatinib
- Cohort A2 DL4A Expansion (Experimental): Lorlatinib will be given at 150 mg orally once daily continuously for 28 days. Patients must be 18 years of age or older at time of enrollment.
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — Lorlatinib will be given orally once daily continuously in 28-day cycles. Lorlatinib will be provided as 5 mg or 25 mg tablets.
  Other Names: PF06463922
Drug: Cyclophosphamide — Cyclophosphamide 250mg/m2/day will be administered as a 30 minute IV infusion on days 1-5 of each cycle
  Other Names: Cytoxan
  Arms: Cohort B2 DL3A; Cohort B2 DL4A; Cohort B2 DL4B; Cohort B2 DL5B
Drug: Topotecan — Topotecan 0.75mg/m2/day will be administered as a 30 minute IV infusion immediately following cyclophosphamide on days 1-5 of each cycle
  Other Names: SKF-104864,Hycamtin®
  Arms: Cohort B2 DL3A; Cohort B2 DL4A; Cohort B2 DL4B; Cohort B2 DL5B
Drug: Filgrastim/pegfilgrastim — Filgrastim is to be given with each course beginning 24-48 hours following completion of cyclophosphamide and topotecan and continued through post-nadir count recovery with an ANC > 2000/mm^3 at 5mcg/kg/day. Filgrastim must be discontinued at least 24 hours prior to the start of the next course of therapy.
  Pegfilgrastim (100mcg/kg; 6mg maximum dose) may be substituted and is given one time at 24-48 hours from completion of cyclophosphamide and topotecan.
  Arms: Cohort B2 DL3A; Cohort B2 DL4A; Cohort B2 DL4B; Cohort B2 DL5B

SUMMARY:
Lorlatinib is a novel inhibitor across ALK variants, including those resistant to crizotinib. In this first pediatric phase 1 trial of lorlatinib, the drug will be utilized as a single agent and in combination with chemotherapy in patients with relapsed/refractory neuroblastoma. The dose escalation phase of this study (Cohort A1) uses a traditional Phase I 3+3 design. Once a recommended phase 2 pediatric dose is identified, an expansion cohort of 6 patients (Cohort B1), within which ALKi naïve patients will be prioritized, will be initiated. Parallel cohorts will be initiated in adults or patients with large BSA (Cohort A2) and in combination with chemotherapy upon establishing RP2D (Cohort B2).

DETAILED DESCRIPTION:
Lorlatinib is a novel inhibitor across ALK variants, including those resistant to crizotinib. An adult phase 1 study established an RP2D of 100mg QD for lorlatinib. In this first pediatric phase 1 trial of lorlatinib, the drug will be utilized as a single agent and in combination with chemotherapy in patients with relapsed/refractory neuroblastoma. The dose escalation phase of this study (Cohort A1) uses a traditional Phase I 3+3 design. Once a recommended phase 2 pediatric dose is identified, an expansion cohort of 6 patients (Cohort B1), within which ALKi naïve patients will be prioritized, will be initiated. Parallel cohorts will be initiated in adults or patients with large BSA (Cohort A2) and in combination with chemotherapy upon establishing RP2D (Cohort B2).

Lorlatinib will be administered orally via tablets or via oral dispersion if patient is unable to swallow tablets whole

All patients will participate in mandatory pharmacokinetic testing.

ELIGIBILITY:
Inclusion Criteria:

1) Patients are required to have an activating ALK aberration in their tumor detected by certified assay (i.e. CLIA in the US.) prior to registration. The report from this test is required to be submitted for eligibility. Patients with at least one of the following genetic features in their tumor will be considered to have an activating ALK aberration:

1. An ALK activating mutation; 2. ALK amplification (> 10 signals of the ALK gene); 3. Presence of any ALK fusion protein that arises from a chromosomal translocation 2) Patients must have a diagnosis of neuroblastoma either by histologic verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines.

3) Patients must have a history of high-risk neuroblastoma according to COG risk classification at the time of study registration. Patients who were initially considered low or intermediate-risk, but then reclassified as high-risk are also eligible.

4) All patients must have at least one of the following

a) Recurrent/progressive disease: after the diagnosis of high risk neuroblastoma at any time prior to enrollment regardless of response to frontline therapy b) No prior history of recurrent/progressive disease since the diagnosis of high risk neuroblastoma b1) Refractory disease- a best overall response of no response/stable disease since diagnosis of high risk neuroblastoma and at least 4 cycles of induction therapy. No prior history of recurrent/progressive disease since the diagnosis of high risk neuroblastoma.

b2) Persistent disease- a best overall response of no partial response since diagnosis of high risk neuroblastoma and at least 4 cycles of induction therapy. No prior history of recurrent/progressive disease since the diagnosis of high risk neuroblastoma.

5) Patients must have at least ONE of the following (lesions may have received prior radiation therapy as long as they meet the other criteria listed below):

1. For recurrent/progressive or refractory disease, at least one MIBG avid bone site.
2. For persistent disease, if a patient has 3 or more MIBG avid lesions, then no biopsy is required. If a patients has only 1 or 2 MIBG avid bone lesion sites then biopsy confirmation of neuroblastoma or ganglioneuroblastoma in at least one MIBG avid site present at the time of enrollment is required to be obtained at any time point prior to enrollment.
3. For MIBG non-avid tumors, patients must have at least one FDG avid site and a biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma at any time prior to enrollment from at least one FDG-avid site.

   6) Any amount of neuroblastoma tumor cells in the bone marrow done at the time of study enrollment based on routine morphology with or without immunocytochemistry in at least one sample from bilateral aspirates and biopsies.

   7) At least one soft tissue lesion that meets criteria for a TARGET lesion as defined by:

<!-- -->

1. SIZE: Lesion can be accurately measured in at least one dimension with a longest diameter ≥ 10 mm, or for lymph nodes ≥ 15 mm on short axis. Lesions meeting size criteria will be considered measurable.
2. In addition to size, a lesion needs to meet one of the following criteria except for patients with parenchymal CNS lesions which only need to meet size criteria:

   b1) MIBG avid. For patients with recurrent/progressive or refractory disease, no biopsy is required. For patients with persistent disease only: If a patient has only 1 or 2 MIBG avid lesions sites, then biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma in at least one MIBG avid site present at time of enrollment is required to be obtained. If a patient has 3 or more MIBG avid lesions, then no biopsy is required.

   b2) MIBG non avid tumors: Patients must have at least one FDG avid site and biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma in at least one FDG-PET avid site present at the time of enrollment.

   8) At least one non-target soft tissue lesion that is not measurable, but had a biopsy positive for neuroblastoma and/or ganglioneuroblastoma or is MIBG avid at any time prior to enrollment.

   9) Patients must have a life expectancy of at least 12 weeks and a Lansky (≤16 years) or Karnofsky (>16 years) score of at least 50.

   10) Prior Therapy
   1. Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to study registration.
   2. Patients must not have received the therapies indicated below after disease evaluation or within the specified time period prior to registration on this study as follows:

   1. Myelosuppressive chemotherapy: must not have received within 2 weeks prior to registration.

   2. Biologic anti-neoplastics- agents not known to be associated with reduced platelet or ANC counts (including retinoids): must not have received within 7 days prior to registration.

   3. Monoclonal antibodies: must have received last dose at least 7 days or 3 half-lives whichever is longer, but no longer than 30 days (with recovery of any associated toxicities), prior to protocol therapy.

   4. Cellular Therapy (e.g. modified T cells, NK cells, dentritic cells etc.): must not have received within 3 weeks and resolution of all toxicities.

   5. Radiation: must not have received small port radiation within 7 days prior to registration.

   6. Hematopoietic Stem Cell Transplant: 7. IVIG 11) All patients must have adequate organ function defined as:

   - Hematological Function:

   1. Absolute Phagocyte count (APC= neutrophils and monocytes): ≥ 1000/µL

   2. Absolute Neutrophil count: ≥750/µL

   3. Absolute Lymphocyte count ≥ 500/µL

   4. Platelet count: ≥ 50,000/µL (A1, A2, and B1); ≥ 75,000/µL (B2), transfusion independent (no platelet transfusions within 1 week)

   5. Hemoglobin ≥ 10 g/dL (may transfuse)

   6. Patients with known bone marrow metastatic disease will be eligible for study as long as they meet hematologic function criteria above.

   - Renal Function: Age-adjusted serum creatinine ≤ to 1.5 x normal for age/gender OR creatinine clearance or GFR greater than or equal to 60 cc/min/1.73m2

   - Liver Function: Total bilirubin ≤ 1.5 x normal for age, AND SGPT (ALT) 135 and SGOT (AST) ≤ 3 x upper limit of normal. Sinusoidal obstruction syndrome (SOS) if present, must be stable or improving clinically

   - Cardiac Function: Normal ejection fraction documented by either echocardiogram or radionuclide MUGA evaluation OR Normal fractional shortening documented by echocardiogram

   - Pulmonary Function: No dyspnea at rest, no oxygen requirement.
   * Neuropsychological Function: Patients must exhibit ≤ grade 1 as defined by CTCAE V4 of nervous system disorders and psychiatric disorders 12) Reproductive Status: All post-menarchal females must have a negative beta-HCG. Males and females of reproductive age and childbearing potential must use effective contraception for the duration of their participation.

     13) Patients with other ongoing serious medical issues must be approved by the study chair prior to registration.

     14) Prior ALK inhibitor treatment- patients must not have been previously treated with lorlatinib. Prior therapy with other ALK inhibitors is allowed.

     15) Concomitant Therapy Restrictions:
     1. Patients may not receive any other anti-cancer agents or radiotherapy while on protocol therapy.
     2. Patient must not be receiving chronic systemic corticosteroids at doses greater than physiologic dosing (inhaled corticosteroids acceptable)
     3. CYP34A inhibitors
     4. CYP34A inducers
     5. CYP34A substrates

   Exclusion Criteria:

   - Pregnancy, breast feeding, or unwillingness to use effective contraception during the study.
   * Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
   * Patients with disease of any major organ system that would compromise their ability to withstand therapy.
   * Patients who have received prior allogeneic stem cell transplant
   * Patients who are on hemodialysis.
   * Patients with an active or uncontrolled infection.
   * Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C.
   * Patient with known history of acute or chronic severe psychiatric disorders
   * Patient with current history of suicidal ideation and history of suicide attempt in their lifetime
   * Patient declines participation in NANT 2004-05, the NANT Biology Study

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yael Mosse, MD, Study Chair — Children's Hospital of Philadelphia
Locations (13):
- United States (10):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children Hospital of Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Chicago, Comer Children's Hospital, Chicago, Illinois
  - Childrens Hospital Boston, Dana-Farber Cancer Institute., Boston, Massachusetts
  - C.S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Healthcare System, Fort Worth, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada
- Institut Curie, Paris, Cedex, France
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goldsmith KC, Park JR, Kayser K, Malvar J, Chi YY, Groshen SG, Villablanca JG, Krytska K, Lai LM, Acharya PT, Goodarzian F, Pawel B, Shimada H, Ghazarian S, States L, Marshall L, Chesler L, Granger M, Desai AV, Mody R, Morgenstern DA, Shusterman S, Macy ME, Pinto N, Schleiermacher G, Vo K, Thurm HC, Chen J, Liyanage M, Peltz G, Matthay KK, Berko ER, Maris JM, Marachelian A, Mosse YP. Lorlatinib with or without chemotherapy in ALK-driven refractory/relapsed neuroblastoma: phase 1 trial results. Nat Med. 2023 May;29(5):1092-1102. doi: 10.1038/s41591-023-02297-5. Epub 2023 Apr 3. PMID 37012551
- [Derived] Baranowska-Kortylewicz J, Kortylewicz ZP, McIntyre EM, Sharp JG, Coulter DW. Multifarious Functions of Butyrylcholinesterase in Neuroblastoma: Impact of BCHE Deletion on the Neuroblastoma Growth In Vitro and In Vivo. J Pediatr Hematol Oncol. 2022 Aug 1;44(6):293-304. doi: 10.1097/MPH.0000000000002285. Epub 2021 Sep 6. PMID 34486544

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort B2 DL4B: Lorlatinib will be given orally once daily continuously for 28 days at 95mg/m2/dose. Lorlatinib should be administered at least one hour prior to conventional chemotherapy (Cyclophosphamide and Topotecan) on days 1-5 of each cycle. Patients must be under 18 years of age at time of enrollment.
  Lorlatinib: Lorlatinib will be given orally once daily continuously in 28-day cycles. Lorlatinib will be provided as 5 mg or 25 mg tablets.
  Cyclophosphamide: Cyclophosphamide 250mg/m2/day will be administered as a 30 minute IV infusion on days 1-5 of each cycle
  Topotecan: Topotecan 0.75mg/m2/day will be administered as a 30 minute IV infusion immediately following cyclophosphamide on days 1-5 of each cycle
  Filgrastim/pegfilgrastim: Filgrastim is to be given with each course beginning 24-48 hours following completion of cyclophosphamide and topotecan and continued through post-nadir count recovery with an ANC > 2000/mm^3 at 5mcg/kg/day. Filgrastim must be discontinued at least 24 hours prior to the start of the next course of therapy.
  Pegfilgrastim (100mcg/kg; 6mg maximum dose) may be substituted and is given one time at 24-48 hours from completion of cyclophosphamide and topotecan.
- Cohort B2 DL5B: Lorlatinib will be given orally once daily continuously for 28 days at 115mg/m2/dose. Lorlatinib should be administered at least one hour prior to conventional chemotherapy (Cyclophosphamide and Topotecan) on days 1-5 of each cycle. Patients must be under 18 years of age at time of enrollment.
  Lorlatinib: Lorlatinib will be given orally once daily continuously in 28-day cycles. Lorlatinib will be provided as 5 mg or 25 mg tablets.
  Cyclophosphamide: Cyclophosphamide 250mg/m2/day will be administered as a 30 minute IV infusion on days 1-5 of each cycle
  Topotecan: Topotecan 0.75mg/m2/day will be administered as a 30 minute IV infusion immediately following cyclophosphamide on days 1-5 of each cycle
  Filgrastim/pegfilgrastim: Filgrastim is to be given with each course beginning 24-48 hours following completion of cyclophosphamide and topotecan and continued through post-nadir count recovery with an ANC > 2000/mm^3 at 5mcg/kg/day. Filgrastim must be discontinued at least 24 hours prior to the start of the next course of therapy.
  Pegfilgrastim (100mcg/kg; 6mg maximum dose) may be substituted and is given one time at 24-48 hours from completion of cyclophosphamide and topotecan.
- Cohort B2 DL3A: Lorlatinib will be given orally once daily continuously for 28 days at 100mg/day. Lorlatinib should be administered at least one hour prior to conventional chemotherapy (Cyclophosphamide and Topotecan) on days 1-5 of each cycle. Patients must be 18 years of age or older at time of enrollment.
  Lorlatinib: Lorlatinib will be given orally once daily continuously in 28-day cycles. Lorlatinib will be provided as 5 mg or 25 mg tablets.
  Cyclophosphamide: Cyclophosphamide 250mg/m2/day will be administered as a 30 minute IV infusion on days 1-5 of each cycle
  Topotecan: Topotecan 0.75mg/m2/day will be administered as a 30 minute IV infusion immediately following cyclophosphamide on days 1-5 of each cycle
  Filgrastim/pegfilgrastim: Filgrastim is to be given with each course beginning 24-48 hours following completion of cyclophosphamide and topotecan and continued through post-nadir count recovery with an ANC > 2000/mm^3 at 5mcg/kg/day. Filgrastim must be discontinued at least 24 hours prior to the start of the next course of therapy.
  Pegfilgrastim (100mcg/kg; 6mg maximum dose) may be substituted and is given one time at 24-48 hours from completion of cyclophosphamide and topotecan.
- Cohort B2 DL4A: Lorlatinib will be given orally once daily continuously for 28 days at 150mg/day. Lorlatinib should be administered at least one hour prior to conventional chemotherapy (Cyclophosphamide and Topotecan) on days 1-5 of each cycle. Patients must be 18 years of age or older at time of enrollment.
  Lorlatinib: Lorlatinib will be given orally once daily continuously in 28-day cycles. Lorlatinib will be provided as 5 mg or 25 mg tablets.
  Cyclophosphamide: Cyclophosphamide 250mg/m2/day will be administered as a 30 minute IV infusion on days 1-5 of each cycle
  Topotecan: Topotecan 0.75mg/m2/day will be administered as a 30 minute IV infusion immediately following cyclophosphamide on days 1-5 of each cycle
  Filgrastim/pegfilgrastim: Filgrastim is to be given with each course beginning 24-48 hours following completion of cyclophosphamide and topotecan and continued through post-nadir count recovery with an ANC > 2000/mm^3 at 5mcg/kg/day. Filgrastim must be discontinued at least 24 hours prior to the start of the next course of therapy.
  Pegfilgrastim (100mcg/kg; 6mg maximum dose) may be substituted and is given one time at 24-48 hours from completion of cyclophosphamide and topotecan.
Period: Overall Study
Arm/Group | Cohort A1 DL1 | Cohort A1 DL2 | Cohort A1 DL3 | Cohort A1 DL4 | Cohort A1 DL5 | Cohort A2 DL 3A | Cohort A2 DL4A | Cohort A2 DL4A Expansion | Cohort B1 DL5 | Cohort B2 DL4B | Cohort B2 DL5B | Cohort B2 DL3A | Cohort B2 DL4A
Started | 3 | 3 | 3 | 10 | 6 | 6 | 6 | 4 | 6 | 3 | 13 | 1 | 1
Completed | 2 | 1 | 1 | 4 | 5 | 4 | 6 | 3 | 5 | 2 | 9 | 1 | 1
Not Completed | 1 | 2 | 2 | 6 | 1 | 2 | 0 | 1 | 1 | 1 | 4 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression or Relapse | 1 | 2 | 2 | 5 | 1 | 1 | 0 | 0 | 0 | 1 | 4 | 0 | 0
Not completed — Ineligible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 65 patients are included in the initial participant flow as 65 patients were enrolled on this protocol. However, 1 patient was determined to be ineligible prior to start of protocol therapy. The 64 patients included in the baseline analysis population represent all eligible enrolled patients on this protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A1 DL1 | Cohort A1 DL2 | Cohort A1 DL3 | Cohort A1 DL4 | Cohort A1 DL5 | Cohort A2 DL 3A | Cohort A2 DL4A | Cohort A2 DL4A Expansion | Cohort B1 DL5 | Cohort B2 DL4B | Cohort B2 DL5B | Cohort B2 DL3A | Cohort B2 DL4A | Total
Number analyzed (Participants) | 3 | 3 | 3 | 10 | 6 | 6 | 6 | 4 | 5 | 3 | 13 | 1 | 1 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 3 | 10 | 6 | 0 | 2 | 0 | 5 | 3 | 13 | 0 | 0 | 48
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 6 | 4 | 4 | 0 | 0 | 0 | 1 | 1 | 16
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 6 | 3 | 4 | 3 | 3 | 2 | 1 | 7 | 1 | 1 | 35
  Male | 1 | 1 | 3 | 4 | 3 | 2 | 3 | 1 | 3 | 2 | 6 | 0 | 0 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 3 | 2 | 2 | 9 | 6 | 5 | 6 | 2 | 5 | 3 | 11 | 1 | 1 | 56
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 5
  White | 3 | 2 | 2 | 8 | 3 | 5 | 6 | 3 | 1 | 2 | 8 | 1 | 1 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 4 | 0 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: MTD/RP2D Determination A1
Description: Proportion of patients with course 1 DLT and/or course 2 neuropsychological DLT in cohort A1
Time Frame: All toxicities from enrollment until completion of course 2 (Day 56)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1 DL1 | Cohort A1 DL2 | Cohort A1 DL3 | Cohort A1 DL4 | Cohort A1 DL5
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 6
Participants | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: MTD/RP2D Determination A2
Description: Proportion of patients with course 1 DLT and/or course 2 neuropsychological DLT in cohort A2
Time Frame: All toxicities from enrollment until completion of course 2 (Day 56)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A2 DL 3A | Cohort A2 DL4A | Cohort A2 DL4A Expansion
Number analyzed (Participants) | 6 | 6 | 4
Participants | 0 | 1 | 2

3. Primary Outcome: MTD/RP2D Determination B2
Description: Proportion of patients with course 1 DLT in cohort B2
Time Frame: All toxicities from enrollment until completion of course 1 (Day 28)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B2 DL4B | Cohort B2 DL5B | Cohort B2 DL3A | Cohort B2 DL4A
Number analyzed (Participants) | 3 | 12 | 1 | 1
Participants | 0 | 1 | 0 | 0

4. Primary Outcome: Describe Non-Hematological Toxicities (A1 and B1)
Description: Proportion of patients with any grade 3 or greater non-hematological toxicities on any course in A1 and B1
Time Frame: All toxicities from enrollment through 30 days following end of protocol therapy, an average of 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1 DL1 | Cohort A1 DL2 | Cohort A1 DL3 | Cohort A1 DL4 | Cohort A1 DL5 | Cohort B1 DL5
Number analyzed (Participants) | 3 | 3 | 3 | 10 | 6 | 5
Participants | 3 | 2 | 1 | 5 | 6 | 4

5. Primary Outcome: Describe Hematological Toxicities (A1 and B1)
Description: Proportion of patients with any grade 3 or greater hematological toxicities on any course in A1 and B1
Time Frame: All toxicities from enrollment through 30 days following end of protocol therapy, an average of 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1 DL1 | Cohort A1 DL2 | Cohort A1 DL3 | Cohort A1 DL4 | Cohort A1 DL5 | Cohort B1 DL5
Number analyzed (Participants) | 3 | 3 | 3 | 10 | 6 | 5
Participants | 0 | 0 | 0 | 5 | 2 | 1

6. Primary Outcome: Describe Non-Hematological Toxicities (A2)
Description: Proportion of patients with any grade 3 or greater non-hematological toxicities in A2
Time Frame: All toxicities from enrollment through 30 days following end of protocol therapy, an average of 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A2 DL 3A | Cohort A2 DL4A | Cohort A2 DL4A Expansion
Number analyzed (Participants) | 6 | 6 | 4
Participants | 6 | 4 | 2

7. Primary Outcome: Describe Hematological Toxicities (A2)
Description: Proportion of patients with any grade 3 or greater hematological toxicities in A2
Time Frame: All toxicities from enrollment through 30 days following end of protocol therapy, an average of 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A2 DL 3A | Cohort A2 DL4A | Cohort A2 DL4A Expansion
Number analyzed (Participants) | 6 | 6 | 4
Participants | 3 | 1 | 0

8. Primary Outcome: Describe Non-Hematological Toxicities (B2)
Description: Proportion of patients with any grade 3 or greater non-hematological toxicities in B2
Time Frame: All toxicities from enrollment through 30 days following end of protocol therapy, an average of 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B2 DL4B | Cohort B2 DL5B | Cohort B2 DL3A | Cohort B2 DL4A
Number analyzed (Participants) | 3 | 13 | 1 | 1
Participants | 3 | 12 | 1 | 1

9. Primary Outcome: Describe Hematological Toxicities (B2)
Description: Proportion of patients with any grade 3 or greater hematological toxicities in B2
Time Frame: All toxicities from enrollment through 30 days following end of protocol therapy, an average of 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B2 DL4B | Cohort B2 DL5B | Cohort B2 DL3A | Cohort B2 DL4A
Number analyzed (Participants) | 3 | 13 | 1 | 1
Participants | 3 | 12 | 1 | 1

10. Secondary Outcome: Pharmacokinetics A1 and B1-Steady State AUC
Description: Steady State AUC for lorlatinib in patients in cohort A1 and B1
Time Frame: Day 1 through Day 15 (0, 1, 2, 24, 360, 361, 362, 364, 366 hours post-initial dose)
Population: No AUCtau is included for patients in Cohort B1DL5 as they do not have the sufficient samples at the necessary time points to calculate a terminal half-life so any estimation would not be reliable.
Measure: Median (Full Range); unit: hours*ng/mL
Arm/Group | Cohort A1 DL1 | Cohort A1 DL2 | Cohort A1 DL3 | Cohort A1 DL4 | Cohort A1 DL5 | Cohort B1 DL5
Number analyzed (Participants) | 2 | 1 | 1 | 6 | 3 | 1
hours*ng/mL | 1872 [1074.93 to 2669.08] | 2663.49 [2663.49 to 2663.49] | 2084.81 [2084.81 to 2084.81] | 7431.06 [3021.81 to 8906.31] | 5655.05 [4724.92 to 10910.87] | NA [NA to NA] — No AUCtau is included for patients in Cohort B1DL5 as they do not have the sufficient samples at the necessary time points to calculate a terminal half-life so any estimation would not be reliable.

11. Secondary Outcome: Pharmacokinetics A2-Steady State AUC
Description: Steady State AUC for lorlatinib in patients in cohort A2
Time Frame: Day 1 through Day 15 (0, 1, 2, 24, 360, 361, 362, 364, 366 hours post-initial dose)
Measure: Median (Full Range); unit: hours*ng/mL
Arm/Group | Cohort A2 DL 3A | Cohort A2 DL4A | Cohort A2 DL4A Expansion
Number analyzed (Participants) | 2 | 3 | 3
hours*ng/mL | 9217.85 [7267.6 to 11168.1] | 4492.92 [3993.55 to 5139] | 5383.5 [4629.88 to 5747.95]

12. Secondary Outcome: Pharmacokinetics B2-Steady State AUC
Description: Steady State AUC for lorlatinib in patients in cohort B2
Time Frame: Day 1 through Day 15 (0, 1, 2, 24, 360, 361, 362, 364, 366 hours post-initial dose)
Population: No AUCtau is included for patients in Cohort B2 DL4B or Cohort B2 DL3A as they do not have the sufficient samples at the necessary time points to calculate a terminal half-life so any estimation would not be reliable.
Measure: Median (Full Range); unit: hours*ng/mL
Arm/Group | Cohort B2 DL4B | Cohort B2 DL5B | Cohort B2 DL3A | Cohort B2 DL4A
Number analyzed (Participants) | 2 | 7 | 1 | 1
hours*ng/mL | NA [NA to NA] — No AUCtau is included for patients in Cohort B2 DL4B as they do not have the sufficient samples at the necessary time points to calculate a terminal half-life so any estimation would not be reliable. | 6310.38 [4695.62 to 14106.75] | NA [NA to NA] — No AUCtau is included for patients in Cohort B2 DL3A as they do not have the sufficient samples at the necessary time points to calculate a terminal half-life so any estimation would not be reliable. | 7594.16 [7594.16 to 7594.16]

13. Secondary Outcome: Overall Response A1 and B1
Description: Proportion of patients evaluable for response with a best overall response of CR/CR-MD/PR for patients in cohort A1 and B1
Time Frame: From Day 1 of protocol therapy through 30 days following end of protocol therapy, an average of 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1 DL1 | Cohort A1 DL2 | Cohort A1 DL3 | Cohort A1 DL4 | Cohort A1 DL5 | Cohort B1 DL5
Number analyzed (Participants) | 3 | 3 | 3 | 9 | 6 | 5
Participants | 1 | 0 | 0 | 0 | 2 | 2

14. Secondary Outcome: Overall Response A2
Description: Proportion of patients evaluable for response with a best overall response of CR/CR-MD/PR for patients in cohort A2
Time Frame: From Day 1 of protocol therapy through 30 days following end of protocol therapy, an average of 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A2 DL 3A | Cohort A2 DL4A | Cohort A2 DL4A Expansion
Number analyzed (Participants) | 6 | 6 | 4
Participants | 2 | 3 | 2

15. Secondary Outcome: Overall Response B2
Description: Proportion of patients evaluable for response with a best overall response of CR/CR-MD/PR for patients in cohort B2
Time Frame: From Day 1 of protocol therapy through 30 days following end of protocol therapy, an average of 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B2 DL4B | Cohort B2 DL5B | Cohort B2 DL3A | Cohort B2 DL4A
Number analyzed (Participants) | 3 | 12 | 1 | 1
Participants | 1 | 5 | 1 | 1

16. Secondary Outcome: Pharmacokinetics A1 and B1-Cmax
Description: Cmax for lorlatinib in patients in cohort A1 and B1
Time Frame: Day 15
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort A1 DL1 | Cohort A1 DL2 | Cohort A1 DL3 | Cohort A1 DL4 | Cohort A1 DL5 | Cohort B1 DL5
Number analyzed (Participants) | 3 | 3 | 3 | 9 | 6 | 1
ng/mL | 287 [243 to 639] | 558 [343 to 623] | 659 [609 to 670] | 1100 [590 to 1880] | 1280 [708 to 2090] | 1800 [1800 to 1800]

17. Secondary Outcome: Pharmacokinetics A2-Cmax
Description: Cmax for lorlatinib in patients in cohort A2
Time Frame: Day 15
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort A2 DL 3A | Cohort A2 DL4A | Cohort A2 DL4A Expansion
Number analyzed (Participants) | 5 | 6 | 4
ng/mL | 569 [341 to 1830] | 710 [502 to 912] | 878.5 [602 to 1100]

18. Secondary Outcome: Pharmacokinetics B2-Cmax
Description: Cmax for lorlatinib in patients in cohort B2
Time Frame: Day 15
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort B2 DL4B | Cohort B2 DL5B | Cohort B2 DL3A | Cohort B2 DL4A
Number analyzed (Participants) | 2 | 11 | 1 | 1
ng/mL | 823.5 [721 to 926] | 1440 [83 to 3340] | 526 [526 to 526] | 1490 [1490 to 1490]

ADVERSE EVENTS:
Time Frame: Timeframe from enrollment through 30 days following end of protocol therapy, an average of 10 months
Arm/Group | Cohort A1 DL1 | Cohort A1 DL2 | Cohort A1 DL3 | Cohort A1 DL4 | Cohort A1 DL5 | Cohort A2 DL 3A | Cohort A2 DL4A | Cohort A2 DL4A Expansion | Cohort B1 DL5 | Cohort B2 DL4B | Cohort B2 DL5B | Cohort B2 DL3A | Cohort B2 DL4A
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/3 | 2/3 | 9/10 | 3/6 | 4/6 | 2/6 | 0/4 | 3/5 | 2/3 | 7/13 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 0/3 | 3/10 | 2/6 | 4/6 | 3/6 | 1/4 | 3/5 | 3/3 | 10/13 | 1/1 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 9/10 | 6/6 | 6/6 | 6/6 | 4/4 | 5/5 | 3/3 | 12/13 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A1 DL1 (N=3) | Cohort A1 DL2 (N=3) | Cohort A1 DL3 (N=3) | Cohort A1 DL4 (N=10) | Cohort A1 DL5 (N=6) | Cohort A2 DL 3A (N=6) | Cohort A2 DL4A (N=6) | Cohort A2 DL4A Expansion (N=4) | Cohort B1 DL5 (N=5) | Cohort B2 DL4B (N=3) | Cohort B2 DL5B (N=13) | Cohort B2 DL3A (N=1) | Cohort B2 DL4A (N=1)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 1 | 1
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1
Flu like symptoms (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TRANSFUSION-ASSOCIATED CIRCULATORY OVERLOAD (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
BILIARY OBSTRUCTION (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID 19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 0
Flu like symptoms (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholesterol high (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PAPILLARY THYROID CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A1 DL1 (N=3) | Cohort A1 DL2 (N=3) | Cohort A1 DL3 (N=3) | Cohort A1 DL4 (N=10) | Cohort A1 DL5 (N=6) | Cohort A2 DL 3A (N=6) | Cohort A2 DL4A (N=6) | Cohort A2 DL4A Expansion (N=4) | Cohort B1 DL5 (N=5) | Cohort B2 DL4B (N=3) | Cohort B2 DL5B (N=13) | Cohort B2 DL3A (N=1) | Cohort B2 DL4A (N=1)
Anemia (Blood and lymphatic system disorders) | 1 | 3 | 1 | 7 | 3 | 4 | 4 | 2 | 3 | 3 | 12 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 2 | 1 | 5 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABNORMAL EYE MOVEMENTS (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid function disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SUBCONJUNCTIVAL HEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ANAL FISSURE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 1 | 1 | 0 | 2 | 1 | 1 | 5 | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 3 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 2 | 3 | 5 | 3 | 2 | 2 | 2 | 3 | 7 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 4 | 1 | 3 | 2 | 3 | 1 | 1 | 5 | 0 | 1
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 5 | 1 | 4 | 3 | 2 | 2 | 1 | 7 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Edema face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Edema limbs (General disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 4 | 2 | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 4 | 1 | 4 | 1 | 0 | 1 | 2 | 8 | 1 | 0
Fever (General disorders) | 0 | 2 | 1 | 4 | 1 | 2 | 0 | 0 | 2 | 2 | 6 | 1 | 1
Flu like symptoms (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Localized edema (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pain (General disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 3 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ASTROVIRUS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bladder infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
COVID 19 (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 4 | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervicitis infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flu like symptoms (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papulopustular rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 2 | 1 | 3 | 1 | 2 | 1 | 1 | 2 | 0 | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulval infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 3 | 2 | 6 | 3 | 4 | 5 | 2 | 4 | 1 | 6 | 1 | 1
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 3 | 2 | 3 | 3 | 2 | 5 | 2 | 8 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 2 | 7 | 3 | 6 | 6 | 2 | 5 | 2 | 6 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholesterol high (Investigations) | 3 | 3 | 3 | 5 | 5 | 6 | 6 | 3 | 5 | 2 | 12 | 1 | 1
Creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 2 | 1 | 3 | 0 | 1 | 0 | 5 | 1 | 0
ELEVATED CRP (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ELEVATED SED RATE (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
GGT increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
HYPERPHOSPHATEMIA (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Hemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
INCREASED UREA (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
LDH INCREASE (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 5 | 1 | 5 | 1 | 1 | 0 | 3 | 11 | 1 | 1
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
NAIL CHANGES (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
NEUTROPHIL COUNT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 2 | 4 | 1 | 0 | 0 | 2 | 3 | 12 | 1 | 1
Pancreatic enzymes decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 2 | 2 | 3 | 4 | 5 | 4 | 1 | 1 | 3 | 12 | 1 | 1
Weight gain (Investigations) | 3 | 3 | 3 | 6 | 5 | 6 | 6 | 3 | 4 | 1 | 9 | 1 | 1
Weight loss (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 0 | 1 | 1 | 3 | 4 | 3 | 2 | 0 | 0 | 3 | 12 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 6 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 3 | 1 | 3 | 2 | 2 | 3 | 2 | 5 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 2 | 2 | 5 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 | 3 | 3 | 8 | 6 | 6 | 6 | 3 | 4 | 2 | 12 | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 5 | 1 | 1 | 0 | 0 | 1 | 1 | 4 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 3 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 5 | 1 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 1 | 3 | 0 | 1 | 1 | 0 | 4 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 2 | 2 | 0 | 1 | 2 | 0 | 4 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0
INCREASED APPETITE (Metabolism and nutrition disorders) | 2 | 2 | 2 | 3 | 3 | 2 | 4 | 2 | 0 | 0 | 3 | 1 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LDL DIRECT INCREASED (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CRAMPS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PATELLAR SUBFIXATION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PAPILLARY THYROID CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 2 | 2 | 1 | 1 | 0 | 0
Concentration impairment (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 3 | 3 | 2 | 2 | 0 | 3 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 4 | 2 | 3 | 3 | 4 | 0 | 1 | 4 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 3 | 4 | 2 | 0 | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
STAMMERING (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
STUTTERING (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 3 | 2 | 2 | 2 | 1 | 1 | 3 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 3 | 5 | 2 | 2 | 0 | 0 | 4 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 2 | 3 | 1 | 1 | 1 | 0 | 2 | 0 | 1
Euphoria (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
REPORT OF FEELING "EMOTIONALLY NUMB" (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 3 | 0 | 2 | 1 | 1 | 0 | 2 | 5 | 1 | 0
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
LEFT HYDROURETER (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NOCTURNAL ENURESIS (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Irregular menstruation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Premature menopause (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 4 | 3 | 4 | 0 | 2 | 3 | 1 | 6 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 2 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 3 | 3 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 5 | 1 | 0
Body odor (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ECCHYMOTIC NODULE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HERPES SIMPLEX REACTIVATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SKIN REACTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 3 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT03107988/Prot_SAP_ICF_000.pdf